CLINICAL TRIAL: NCT04232956
Title: Is Invasive Pulmonary Aspergillosis a Common Complication of Severe Influenza ?
Brief Title: Invasive Pulmonary Aspergillosis and Severe Influenza
Acronym: ASPERGIGRIPP
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: ASPERGIGRIPP (29BRC18.0069)
Record Dates: First submitted 2018-07-10; First posted 2020-01-18 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Aspergillosis; Influenza; Critical Illness
MeSH Terms: conditions — Aspergillosis; Influenza, Human; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Invasive pulmonary aspergillosis (IPA) has been reported in critically ill patients with influenza infection with a highly variable incidence between 1 to 21%. Studies investigating IPA in critically ill patients with influenza infection suffer limitations in their methods. It remains unknown whether patients with influenza are more at risk of IPA than other patients hospitalized in intensive care unit and whether patients with influenza who develop IPA have specific risk factors for this infection.

Our study aims to determine the incidence of IPA in a large multicenter cohort and to identify risk factors for IPA in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Infection with influenza A or B
* Admission to one of the participating sites

Exclusion Criteria:

* age < 18
* patients with invasive pulmonary aspergillosis prior to intensive care admission
* consent withdraw

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients with influenza infection
Sampling Method: Non-Probability Sample
Enrollment: 478 (Actual)
Dates: Start 2018-07-27 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-05 (Actual)

PRIMARY OUTCOMES:
Invasive Pulmonary Aspergillosis | up to 100 days
  incidence of invasive pulmonary aspergillosis

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHRU de Brest, Brest
  - CHR, Morlaix
  - CHU de NANTES, Nantes
  - CHU de Rennes, Rennes

IPD SHARING:
Plan to Share IPD: No